CLINICAL TRIAL: NCT02581644
Title: Evaluation of the Effectiveness of the Belatacept (Nulojix®) Patient Alert Cards in Patients Following Renal Transplantation in European Economic Area Countries
Brief Title: Assessment of Effectiveness of Belatacept Patient Alert Card in Patients Following Renal Transplantation in a Sample of EU Countries
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM103-367
Record Dates: First submitted 2015-09-28; First posted 2015-10-21 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Renal Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients survey: Adult patients treated with belatacept for renal transplantation
- HCP survey: HCP with at least 1 patient taking belatacept
- Retrospective chart review study: Adult patients treated with belatacept for renal transplantation

SUMMARY:
The purpose of the study is to determine a) if the implementation of belatacept patient alert card (PAC) resulted in effective understanding of key safety messages and b) if the degree of understanding of key safety messages is associated with improved clinical and safety outcomes.

DETAILED DESCRIPTION:
3 sub studies: 2 Cross-Sectional and 1 retrospective chart review

ELIGIBILITY:
Inclusion Criteria:

* Patient survey (cohort 1):
* Patients has taken belatacept within the previous 3 months for renal transplantation
* Patient is over 18 years of age
* HCP survey (cohort 2):
* Physician or nurses working in nephrology centers, with at least 1 patient taking belatacept in the previous 6 months for renal transplantation (by prescribing, administering or by follow up)
* Retrospective chart review study (cohort 3):
* Patient survey questionnaire received, Informed Consent Form (ICF) signed (if required)

Exclusion Criteria:

* Patient survey:
* Patient has participated in a clinical trial for their renal condition in the previous 12 months
* Currently an employee of BMS
* HCP survey:
* Physicians or nurse who have recruited patients for the Patient survey
* Currently an employee of BMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Patient enrolled by physicians based in hospital and physician renal units
  Cohort 2: Physicians and nurses based in hospital and physician renal units
  Cohort 3: Patient enrolled by physicians based in hospital and physician renal units
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Patient survey: Proportion of patients treated with belatacept who are aware of the existence of the PAC | At patient enrolment
Patient survey : Proportion of patients treated with belatacept who have received the PAC | At patient enrolment
Patient survey : Proportion of patients who have utilised the PAC, and the extent of its use | At patient enrolment
Patient survey: Levels of patient knowledge and comprehension related to the important identified risks of belatacept treatment | At patient enrolment
Patient survey: HCP-patient communication based on responses to specific questions | At patient enrolment
Patient survey: Proportion of patients with correct responses to behavioral questions | At patient enrolment
Patient survey: Mean scores for correct responses for questions grouped by objectives | At patient enrolment
  Objectives: distribution, awareness, utility, utilization and knowledge
HCP survey: Proportion of HCPs who prescribe or administer belatacept in nephrology centres who are aware of the PAC | Day 1
HCP survey: Proportion of HCPs who have utilised the PAC, and the extent of its use | Day 1
HCP survey: Levels of HCPs' knowledge and comprehension related to the important identified risks of infections and the need to screen for specific infection prior to initiating or administering belatacept | Day 1
  The percentage of HCPs with responses to each question in the HCP questionnaire that would indicate effectiveness of the PAC will be determined: who are aware of the PAC, use the PAC, level of knowledge and comprehension of the risks and mean scores for correct responses
HCP survey: Behavior of HCPs based on responses to behavioral questions | Day 1
HCP survey: Mean total score for correct responses | Day 1
HCP survey: Mean scores for correct responses for questions grouped by objectives | Day 1
  Objectives: distribution, awareness, utility, utilization and knowledge
Retrospective chart review study (clinical outcome study): Proportion of serious infections | Upto 4 years

SECONDARY OUTCOMES:
Major determinants of patients knowledge of the key messages contained in the belatacept PAC based on data collected in the patient questionnaire | At patient enrolment
  Determinants: Age, gender, educational level, number of prescription medications, duration of therapy with belatacept
Major determinants of understanding the key messages contained in the PAC based on data collected in the patient questionnaire | At patient enrolment
  Determinants: Age, gender, educational level, number of prescription medications, duration of therapy with belatacept
Major determinants of implementation regarding the key messages contained in the PAC based on data collected in the patient questionnaire | At patient enrolment
  Determinants: Age, gender, educational level, number of prescription medications, duration of therapy with belatacept
Determinants of Health Care Professional (HCP) understanding and implementation regarding key messages contained in the PAC based on data collected in the patient questionnaire | Day 1
  Determinants: type of HCP, country, age and gender of HCP years in specialty, number of HCPs in the unit, annual number of patients through the unit, number of patients for whom belatacept was prescribed in the previous 12 months, type of practice, type of institution (academic or non-academic), size of town
Retrospective chart review study (clinical outcome study) : proportion of infections leading to discontinuation | Upto 4 years
Retrospective chart review study (clinical outcome study) : mean time from symptom onset of infection to receipt of medical therapy | Upto 4 years
Retrospective chart review study (clinical outcome study) : Mean time to diagnosis of graft rejection by biopsy criteria | Upto 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- Austria (2):
  - Local Institution, Linz
  - Local Institution, Vienna
- France (8):
  - Local Institution, Besançon
  - CHU Brest Hopital La Cavale Blanche, Brest
  - CHU Bordeaux Hopital Pellegrin, Burdeux
  - CHU Clemont Ferrand, Clermont-Ferrand
  - APHP Hopital Henri Mondor, Créteil
  - Local Institution, Le Kremlin-Bicêtre
  - CHU Toulouse Hopital Rangueli, Toulouse
  - CHU Tours Hopital Bretonneau, Tours
- Germany (3):
  - Local Institution, Dresden
  - Local Institution, Kiel
  - UK Mannheim, Mannheim
- Local Institution, Uppsala, Sweden

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx